CLINICAL TRIAL: NCT00973050
Title: Randomized, 1-Way Parallel, Bioequivalence Study of Bicalutamide 50 mg Tablets and Casodex® Administered as 1 x 50 mg Tablet in Healthy Subjects Under Fasting Conditions
Brief Title: Study of Bicalutamide 1 x 50 mg Tablet in Healthy Subjects Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 30062
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
Keywords: Bioequivalence
MeSH Terms: interventions — bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bicalutamide (test) (Experimental): Bicalutamide Tablet, 50 mg
  Interventions: Drug: Bicalutamide
- Casodex® (reference) (Active Comparator): Casodex® Tablet, 50 mg
  Interventions: Drug: Casodex®

INTERVENTIONS:
Drug: Bicalutamide — 50 mg Tablet
  Arms: Bicalutamide (test)
Drug: Casodex® — 50 mg Tabelt
  Arms: Casodex® (reference)

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of bicalutamide 50 mg tablets (test) versus Casodex® (reference) administered as 1 x 50 mg tablet under fasting conditions.

DETAILED DESCRIPTION:
This will be a single center, bioequivalence, open-label, randomized, 1-way parallel study.

According to the BA/BE guidances, a parallel study is acceptable for drugs with a long half-life.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be males, non-smokers, 18 years of age and older.

Exclusion Criteria:

Subjects to whom any of the following applies will be excluded from the study:

* Clinically significant illnesses within 4 weeks of the administration of study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the medical subinvestigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive urine drug screen at screening.
* Positive testing for hepatitis B, hepatitis C or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, or diastolic blood pressure lower than 50 or over 90; or heart rate less than 50 bpm) at screening.
* Subjects with BMI ≥30.0.
* History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than two units of alcohol per day (1 Unit = 150 mL of wine or 360 mL of beer or 45 mL of alcohol 40%).
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PCP) and crack) within 1 year of the screening visit.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the medical subinvestigator, contraindicates the subject's participation in this study.
* History of allergic reactions to bicalutamide or other related drugs.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin; examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin, ketoconazole, MAO inhibitors, neuroleptics, verapamil, quinidine) within 30 days prior to the administration of the study medication.
* Use of an investigational drug or participation in an investigation study within 30 days prior to the administration of the study medication.
* Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug.
* Any clinically significant history or presence of clinically significant neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Any food allergy, intolerance, restriction or special diet that could, in the opinion of the medical subinvestigator, contraindicate the subjects participation in this study.
* A depot injection or an implant of any drug within 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days. Donation or loss of whole blood prior to administration of the study medication as follows:
* Less than 300 mL of whole blood within 30 days or
* 300 mL to 500 mL of whole blood within 45 days or
* more than 500 mL of whole blood within 56 days.
* Positive alcohol breath test at screening.
* Subjects who have used tobacco in any form within the 90 days preceding study drug administration.
* Subjects with a clinically significant history of tuberculosis, epilepsy, asthma, diabetes, psychosis or glaucoma.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-09; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Cmax - Maximum Observed Concentration | Blood samples collected over 72 hour period
AUC0-72: Area under the concentration-time curve from time zero to 72 hours post-dose. | Blood samples collected over 72 hour period

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, MD, Principal Investigator — Anapharm
Locations (1):
- Anapharm Inc., Sainte-Foy, Quebec, Canada